CLINICAL TRIAL: NCT00732043
Title: A 48-Month Extension to the Randomized, Double-blind, Placebo-Controlled Study of the Effects of Pomegranate Extract on Rising Prostate-Specific Antigen Levels in Men Following Primary Therapy for Prostate Cancer
Brief Title: Extension to Study of Effects of Pomegranate Extract on Rising PSA Levels After Primary Therapy for Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Roll International Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GUP-0205-1XX
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate-specific antigen; PSA; pomegranate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pomegranate fruit rind

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Dietary Supplement: pomegranate extract
- 2 (Experimental)
  Interventions: Dietary Supplement: pomegranate juice
- 3 (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: pomegranate extract — 8 oz per day, 48 months
  Arms: 1
Dietary Supplement: pomegranate juice — 8 oz per day, 48 months
  Other Names: PomWonderful
  Arms: 2
Dietary Supplement: placebo — 8 oz per day, 48 months
  Arms: 3

SUMMARY:
High concentrations of anti-oxidants in pomegranate seeds present a potential strategy to delay clinical prostate cancer progression and prolong the interval from primary treatment failure to hormonal ablation. This is a 48 month extension to the double-blind GUP-0205-1 study, to compare the effects of daily consumption of pomegranate liquid extract versus placebo on the absolute prostate-specific antigen (PSA) doubling time at the end of 12, 24, 36 and 48 months in male subjects who rolled-over from the GUP-0205-1 study.

DETAILED DESCRIPTION:
The primary objectives are to compare the effects of daily consumption of pomegranate liquid extract versus placebo on the absolute prostate-specific antigen (PSA) doubling time at the end of 12,24, 36 and 48 months in male subjects who rolled-over from the GUP-0205-1 study. Secondary objectives are to determine the effect of the pomegranate treatment on the change in PSA doubling time from baseline to each 12-month visit, to determine the time to tumor recurrence, to assess the tolerability and toxicity of the pomegranate treatment and to determine the effect of the pomegranate treatment on response rates for positive PSA doubling times and for declining post-treatment PSA levels (negative doubling times).

ELIGIBILITY:
Inclusion Criteria:

* No evidence of disease progression while on any of the three GUP-0205 study products (disease progression defined as > 100% increase in serum PSA [with a minimum value of 1.0 ng/mL]).
* Willingness and ability to sign an informed consent document.
* Agreement with complete abstinence from other commercially available pomegranate products during the course of the study.
* Use of dietary/herbal supplements (e.g., saw palmetto, selenium, etc) is acceptable provided the dose has been stable during the course of the GUP-0205- 1 study.

Exclusion Criteria:

* Significant concomitant medical or psychiatric condition that, in the opinion of the Principal Investigator, would put the subject at risk or compromise the protocol.
* Hormonal therapy, with the exception of neoadjuvant androgen deprivation therapy (ADT) prior to or concurrent with primary therapy. Subjects who underwent neoadjuvant ADT cannot have a serum testosterone of ≤150 ng/mL at study entry.
* Concomitant or antecedent hormonal therapy for rising serum PSA after initial therapy of prostate cancer.
* Subjects unable or unwilling to comply with protocol requirements.
* Prior treatment with experimental drugs, high dose steroids, or with any other cancer treatment within 4 weeks prior to the first dose of study product and for the duration of the study.
* Serum PSA >7.0 ng/mL (assessed at termination of the double-blind study; at any PSA level, the subject will be excluded if determined by the Principal Investigator that the subject's continued participation would not be in their best interest).
* Serum PSA doubling time <13 weeks (assessed at termination of the double-blind study).
* Evidence of metastatic disease on physical examination or on CT or bone scan.
* Use of finasteride, dutasteride at any point since primary therapy or during the study.
* Clinically significant abnormal laboratory value greater than 2 times the upper limit of normal (>2XULN).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-12; Primary Completion 2014-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome variable will be the mean PSA doubling time at the end of 12, 24,36 and 48 months. | 48 months

SECONDARY OUTCOMES:
The mean change in PSA doubling time from baseline to end-of-treatment. | 48 months
Response rates in positive and negative PSA doubling times with a clinically significant positive doubling time is defined as >150% of baseline. | 48 months
Overall efficacy responses categorized as Objective Response, Progressive Disease, Stable Disease. | 48 months
Measures of tolerability (adverse events) and toxicity (clinical chemistries, etc.). | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Allan J Pantuck, MD, Principal Investigator — University of California, Los Angeles; Arie S Belldegrun, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA School of Medicine, Los Angeles, California, United States